CLINICAL TRIAL: NCT04732988
Title: A Dose-block Randomized, Double-blind, Placebo-controlled, Single and Multiple Dosing, Dose-escalation Phase I Clinical Trial to Investigate the Safety, Tolerability, Pharmacokinetic/Pharmacodynamic Characteristics, and Food Effect of HSG4112 After Oral Administration in Healthy and Obese Male Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetic/Pharmacodynamic Characteristics, and Food Effect of HSG4112
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glaceum (Industry)
Collaborators: Seoul National University Hospital (Other); Kyungpook National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSG4112-P1-01
Record Dates: First submitted 2021-01-19; First posted 2021-02-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (17):
- HSG4112 30 mg Single Dose (Experimental): Single oral dosing of HSG4112 30 mg
  Interventions: Drug: HSG4112
- Placebo 30 mg Single Dose (Placebo Comparator): Single oral dosing of Placebo 30 mg
  Interventions: Drug: Placebo
- HSG4112 60 mg Single Dose (Experimental): Single oral dosing of HSG4112 60 mg
  Interventions: Drug: HSG4112
- Placebo 60 mg Single Dose (Placebo Comparator): Single oral dosing of Placebo 60 mg
  Interventions: Drug: Placebo
- HSG4112 120 mg Single Dose (Experimental): Single oral dosing of HSG4112 120 mg
  Interventions: Drug: HSG4112
- Placebo 120 mg Single Dose (Placebo Comparator): Single oral dosing of Placebo 120 mg
  Interventions: Drug: Placebo
- HSG4112 240 mg Single Dose (Fasted) (Experimental): Single oral dosing of HSG4112 240 mg under fasted conditions
  Interventions: Drug: HSG4112
- HSG4112 240 mg Single Dose (Fed) (Experimental): Single oral dosing of HSG4112 240 mg under fed conditions
  Interventions: Drug: HSG4112
- Placebo 240 mg Single Dose (Placebo Comparator): Single oral dosing of Placebo 240 mg
  Interventions: Drug: Placebo
- HSG4112 480 mg Single Dose (Experimental): Single oral dosing of HSG4112 480 mg
  Interventions: Drug: HSG4112
- Placebo 480 mg Single Dose (Placebo Comparator): Single oral dosing of Placebo 480 mg
  Interventions: Drug: Placebo
- HSG4112 720 mg Single Dose (Experimental): Single oral dosing of HSG4112 720 mg
  Interventions: Drug: HSG4112
- Placebo 720 mg Single Dose (Placebo Comparator): Single oral dosing of Placebo 720 mg
  Interventions: Drug: Placebo
- HSG4112 240 mg Multiple Dose (Experimental): Once-daily multiple oral dosing of HSG4112 240 mg for 14 days
  Interventions: Drug: HSG4112
- Placebo 240 mg Multiple Dose (Placebo Comparator): Once-daily multiple oral dosing of Placebo 240 mg for 14 days
  Interventions: Drug: Placebo
- HSG4112 480 mg Multiple Dose (Experimental): Once-daily multiple oral dosing of HSG4112 480 mg for 14 days
  Interventions: Drug: HSG4112
- Placebo 480 mg Multiple Dose (Placebo Comparator): Once-daily multiple oral dosing of Placebo 480 mg for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSG4112 — Once-daily oral administration
  Other Names: 2-(8,8 dimethyl 2,3,4,8,9,10 hexahydropyrano[2,3 f]chromen 3 yl) 5 ethoxyphenol
  Arms: HSG4112 120 mg Single Dose; HSG4112 240 mg Multiple Dose; HSG4112 240 mg Single Dose (Fasted); HSG4112 240 mg Single Dose (Fed); HSG4112 30 mg Single Dose; HSG4112 480 mg Multiple Dose; HSG4112 480 mg Single Dose; HSG4112 60 mg Single Dose; HSG4112 720 mg Single Dose
Drug: Placebo — Once-daily oral administration
  Arms: Placebo 120 mg Single Dose; Placebo 240 mg Multiple Dose; Placebo 240 mg Single Dose; Placebo 30 mg Single Dose; Placebo 480 mg Multiple Dose; Placebo 480 mg Single Dose; Placebo 60 mg Single Dose; Placebo 720 mg Single Dose

SUMMARY:
1. Study Objective: The objective of this phase 1 clinical trial is to evaluate the safety, tolerability, pharmacokinetic/pharmacodynamic characteristics and food effect of HSG4112 after oral administration in healthy male subjects.
2. Study Design and Plan: This study is a dose-block randomized, double-blind, placebo-controlled, single and multiple dosing, dose-escalation phase 1 clinical trial. A unique randomization number will be assigned to each subject deemed eligible to participate in the study based on the inclusion/exclusion criteria. Each subject will be randomized to one of the six groups for the single ascending dose (SAD) study or one of the three groups for the multiple ascending dose (MAD) study. Each dose group will consist of ten subjects, and among the ten subjects, eight subjects will be randomized to receive HSG4112 and two subjects will be randomized to receive placebo. The subjects will be studied in a double-blind manner and will receive the investigational product (i.e., HSG4112 or placebo) via once-daily oral administration. The dosing duration for the MAD study is 14 days. When escalating the dose, the Investigator will review all of the available safety data from the preceding dose in a blinded manner to ensure if it is safe to escalate the dose. In order to evaluate safety and tolerability, assessments, such as vital signs, 12-lead electrocardiogram, laboratory test, semen analysis (MAD study only), physical examination, and adverse event monitoring will be performed. Blood samples will be collected to evaluate the pharmacokinetic/pharmacodynamic characteristics of HSG4112.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form approved by the IRB before screening.
2. Males between 19 and 50 years of age at screening.
3. Body mass index (BMI) between 18 and 24.9.

   ☞ BMI (kg/m2) = Body weight (kg) / {Height (m)2}
4. In good health, determined by no clinically significant findings from medical history, physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory test at screening, or subjects who are deemed acceptable by the Investigator regardless of the test results.

Exclusion Criteria:

1. Significant history or clinical manifestation of any hepatic, kidney, neurological, immune, respiratory, endocrine, hematological, neoplastic, or cardiovascular disease, or psychiatric disorder (e.g., mood disorder, obsessive-compulsive disorder).
2. History of stomach or intestinal disorders (e.g., Chrons disease, ulcer) or surgeries - not including appendectomy, hemorrhoidectomy, or herniotomy - which may affect the pharmacokinetic or pharmacodynamic evaluation of the investigational product.
3. Significant history or clinical manifestation of hypersensitivity to any drug compound (e.g., licorice, aspirin, antibiotics).
4. One of more of the following laboratory test results at screening:

   * ALT (SGPT) > 60 IU/L
   * Glucose (fasting) > 110 mg/dL or < 70 mg/dL
   * Testosterone <2.49 ng/mL or > 8.36 ng/mL
5. Systolic blood pressure of < 90 mmHg or > 150 mmHg, or diastolic blood pressure of < 60 mmHg or > 100 mmHg as determined by vital signs monitored after resting in sitting position for at least 3 minutes.
6. History of drug/chemical abuse or tested positive in urine drug screen.
7. Use or intend to use any prescription medications/products or phytotherapeutic/herbal/plant-derived preparations within 14 days prior to dosing, or any nonprescription medications/products (i.e., over-the-counter (OTC) drugs), health products, or vitamins within 7 days prior to dosing, unless deemed acceptable by the Investigator.
8. Participation in any clinical study or bioequivalence study involving administration of an investigational drug, including any study investigating HSG4112, within 6 months prior to dosing (i.e., within 6 months of the last dose from the previous study).
9. Whole blood donation within 2 months prior to dosing, plasma/platelet donation within 1 month prior to dosing, or receipt of blood products within 1 month prior to dosing, or receipt of blood products within 1 month prior to dosing.
10. Alcohol consumption of > 20 units/week (1 unit = 10 g of pure alcohol) or unable to abstain from consuming alcohol during the study period.
11. Smoked within 90 days prior to dosing. However, participation is acceptable if the subject has quit smoking at least 90 days prior to dosing.
12. Smoker. However, participation is acceptable if the subject has quit smoking at least 3 months prior to dosing.
13. Ingestion of grapefruit-containing foods or beverages 24 hours prior to dosing until discharge, or unable to abstain from ingesting such foods or beverages during the same period.
14. Unable to abstain from caffeine-containing foods or beverages (e.g., coffee, tea (e.g., black tea, green tea), soft drinks, coffee milk, energy drinks, sports drinks) during the admission period.
15. Unable or unwilling to use acceptable contraceptive methods during the study period.

    ☞ Acceptable contraceptive methods include:
    * Use of an intrauterine device, which has been proven highly effective, by the subject's spouse/partner.
    * Physical contraception for subject or spouse/partner used with chemical sterilization.
    * Surgical sterilization (e.g., vasectomy, hysterectomy, tubal ligation, salpingectomy) of the subject or the subject's spouse/partner.
16. Subjects who, in the opinion of the Investigator, should not participate in this study based on clinical laboratory test results or other reasons.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 Over Dosing Interval | Hour 0 to 24
  Area under the plasma concentration-time curve of HSG4112 over dosing interval (AUCtau)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to the Last Measurable Point | Hour 0 to 192
  Area under the plasma concentration-time curve from time zero to the last measurable point (AUClast)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to Infinity | Hour 0 to 192
  Area under the plasma concentration-time curve from time zero to infinity (AUCinf)
Pharmacokinetic Assessment by Maximum Plasma Concentration of HSG4112 | Hour 0 to 192
  Maximum plasma concentration of HSG4112 (Cmax)
Pharmacokinetic Assessment by Time to Maximum Observed Plasma Concentration of HSG4112 | Hour 0 to 192
  Time to maximum observed plasma concentration of HSG4112 (Tmax)
Pharmacokinetic Assessment by Half-Life of HSG4112 | Hour 0 to 192
  Half-life of HSG4112 (T1/2)
Pharmacokinetic Assessment by Oral Clearance of HSG4112 | Hour 0 to 192
  Oral clearance of HSG4112 (CL/F)
Pharmacokinetic Assessment by Volume of Distribution of HSG4112 | Hour 0 to 192
  Volume of distribution of HSG4112 (Vd/F)
Safety and Tolerability Assessment by Adverse Event Monitoring | Up to 12 weeks from day of last dosing
  Number of participants with observed adverse events
Safety and Tolerability Assessment by Number of Participants with Change in Vital Signs | Up to 3 weeks from day of last dosing
  Number of participants with clinically significant change in vital signs including blood pressure (mmHg) measured with blood pressure monitor, heart rate (beats per minute) measured with pulse oximeter, and body temperature (degrees Celcius) measured with thermometer
Safety and Tolerability Assessment by Number of Participants with Change in 12-Lead Electrocardiogram | Up to 3 weeks from day of last dosing
  Number of participants with clinically significant change in 12-lead electrocardiogram
Safety and Tolerability Assessment by Number of Participants with Change in Laboratory Test | Up to 3 weeks from day of last dosing
  Number of participants with clinically significant change in laboratory test assessed through hematology, blood biochemistry, urinalysis, and blood coagulation test
Safety and Tolerability Assessment by Number of Patients with Change in Physical Examination | Up to 3 weeks from day of last dosing
  Number of participants with clinically significant change in physical examination
Safety and Tolerability Assessment by Number of Patients with Change in Semen Volume | Up to 12 weeks from day of last dosing
  Pre-to-post examination of semen volume (milliliters) by semen analysis to assess the safety and tolerability of HSG4112
Safety and Tolerability Assessment by Number of Patients with Change in Semen pH | Up to 12 weeks from day of last dosing
  Pre-to-post examination of semen white blood cells (10^3 per microliter) by semen analysis to assess the safety and tolerability of HSG4112
Safety and Tolerability Assessment by Number of Patients with Change in Semen White Blood Cells | Up to 12 weeks from day of last dosing
  Pre-to-post examination of semen white blood cells (10^3 per microliter) by semen analysis to assess the safety and tolerability of HSG4112
Safety and Tolerability Assessment by Number of Patients with Change in Sperm Count | Up to 12 weeks from day of last dosing
  Pre-to-post examination of sperm count (10^6 per milliliter) by semen analysis to assess the safety and tolerability of HSG4112
Safety and Tolerability Assessment by Number of Patients with Change in Sperm Motility | Up to 12 weeks from day of last dosing
  Pre-to-post examination of sperm motility (percent of sperm with normal motility) by semen analysis to assess the safety and tolerability of HSG4112
Safety and Tolerability Assessment by Number of Patients with Change in Sperm Morphology | Up to 12 weeks from day of last dosing
  Pre-to-post examination of sperm morphology (percent of normal sperm) by semen analysis to assess the safety and tolerability of HSG4112

SECONDARY OUTCOMES:
Pharmacodynamic Assessment by Change of Biomarkers | Day 1 and 14 pre-dose
  Measurement of biomarkers including leptin, adiponectin, insulin, C-peptide (connecting peptide), IL6 (interleukin 6), TNF-alpha (tumor necrosis factor alpha), and CCL2 (C-C motif ligand 2) from baseline to day of last dosing will be combined to assess the weight loss effect of HSG4112

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No